CLINICAL TRIAL: NCT02470468
Title: A Phase I/II Study to Evaluate Safety and Efficacy of DCVAC/LuCa Added to Standard First Line ChT With Carboplatin and Paclitaxel +/- Immune Enhancers (Interferon-α and Hydroxychloroquine) vs ChT Alone in Patients With Stage IV NSCLC
Brief Title: Evaluation of Safety and Efficacy of DCVAC/LuCa (Immunotherapy of Lung Cancer) in Patients With Metastatic Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLU01; 2014-003084-37 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Stage IV Non-small Cell Lung Cancer
Keywords: Immunotherapy; Metastatic; NSCLC; Biological; Lung Cancer; Vaccine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — S-1,2-dichlorovinyl-N-acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DCVAC add on to SOC (Experimental): Combination therapy with DCVAC and Standard of Care (Carboplatin, Paclitaxel)
  Interventions: Biological: DCVAC add on to SOC
- DCVAC and immune enhancers add on to SOC (Experimental): Combination therapy with DCVAC, immune enhancers (Interferon-α, Hydroxychloroquine) and Standard of Care (Carboplatin, Paclitaxel)
  Interventions: Biological: DCVAC and immune enhancers add on to SOC
- Standard of Care Chemotherapy (Other): Standard of Care chemotherapy (Carboplatin, Paclitaxel)
  Interventions: Other: Standard of Care Chemotherapy

INTERVENTIONS:
Biological: DCVAC add on to SOC — DCVAC add on to SOC (Carboplatin, Paclitaxel): until progression or intolerance or death
  Arms: DCVAC add on to SOC
Biological: DCVAC and immune enhancers add on to SOC — DCVAC +/- immune enhancers (Interferon-α and Hydroxychloroquine) add on to SOC (Carboplatin, Paclitaxel): until progression or intolerance or death
  Arms: DCVAC and immune enhancers add on to SOC
Other: Standard of Care Chemotherapy — SOC (Carboplatin, Paclitaxel): until progression or intolerance or death
  Arms: Standard of Care Chemotherapy

SUMMARY:
The purpose of the study is to compare efficacy of DCVAC/LuCa + chemotherapy +/- immune enhancers vs. chemotherapy alone in patients with stage IV NSCLC, as measured by progression free survival (PFS).

DETAILED DESCRIPTION:
The purpose of the study is to compare efficacy of DCVAC/LuCa + chemotherapy +/- immune enhancers vs. Standard of Care chemotherapy alone in patients with stage IV NSCLC, as measured by progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) of either adenomatous or squamous cell carcinoma differentiation; mixed tumors will be categorized by the predominant cell type.
2. Advanced NSCLC (stage IV unresectable disease)
3. Patients must have measurable or non-measurable disease
4. Patients (male and female) ≥ 18 years
5. Eastern Cooperative Oncology Group (ECOG) Performance status 0-1 6. Patients must have recovered from toxicity of any prior therapy (e.g. surgery, radiotherapy, or therapy for other diseases than NSCLC). Recovery is defined as less than or equal to grade 2 toxicity according (except alopecia) to NCI CTCAE 7. Laboratory criteria 7.1 Platelet count of at least 100,000/mm3 (100 x 109/L) 7.2 White blood cells (WBC) greater than 4,000/mm3 (4.0 x109/L) 7.3 Hemoglobin (Hb) at least 9g/dL (90 g/L) 7.4 Total bilirubin levels ≤1.5mg/dL (benign hereditary hyper-bilirubinemias, e.g., Gilbert´s syndrome are permitted) 7.5 Serum alanine aminotransferase and aspartate aminotransferase ≤ 5 times the upper limit of normal (ULN) 7.6 Serum creatinine ≤ 1.5 times the upper limit of normal (ULN)

8. Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the treatment plus 3 months.

9. Signed informed consent including patient's ability to comprehend its contents. (Consent to genetic testing is not a condition for participation in the clinical trial)

Exclusion Criteria:

1. Prior chemotherapy for stage IV NSCLC
2. Immunotherapy, monoclonal antibodies received within 4 weeks prior to randomization
3. Patients comorbidities 3.1 Patients who are not indicated for chemotherapy treatment with first line Standard of Care chemotherapy (carboplatin/paclitaxel) 3.2 Active other malignancy than NSCLC 3.3 Known central nervous system (CNS) metastases 3.4 Any disease requiring chronic steroid or immunosuppressive therapy 3.5 HIV positive 3.6 Active hepatitis B (HBV) and/or C (HCV), active syphilis 3.7 Ongoing/active significant infection or other severe medical condition 3.8 Pre-existing thyroid disease unless it can be controlled with conventional treatment 3.9 Clinically significant cardiovascular disease including: 3.9.1 Uncontrolled congestive heart failure 3.9.2 Unstable angina pectoris 3.9.3 Uncontrolled severe cardiac arrhythmia 3.9.4 Myocardial infarction within 6 months prior randomization 3.10 Psychiatric illness/social situations that would limit compliance with study requirements
4. Pregnant or breast feeding women
5. Participation in a clinical trial using experimental therapy within the last 4 weeks prior to randomization
6. Contra indications to treatment with hydroxychloroquine, known G6PD deficiency (anamnestic information, no test necessary) and psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Comparison efficacy of DCVAC/LuCa + chemotherapy +/- immune enhancers vs. chemotherapy alone in patients with stage IV NSCLC, as measured by progression free survival (PFS). | 17 months

SECONDARY OUTCOMES:
Comparison of safety in patients treated with DCVAC/LuCa + chemotherapy +/- immune enhancers vs. chemotherapy alone. (AEs, SAEs, laboratory abnormalities, vital signs) | 17 months
Further comparison of efficacy of DCVAC/LuCa + chemotherapy +/- immune enhancers vs. chemotherapy alone, as measured by objective response rate and duration of response (per RECIST 1.1). | 17 months
Further comparison of efficacy of DCVAC/LuCa + chemotherapy +/- immune enhancers vs. chemotherapy alone, as measured by overall survival. | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Scheiner, Study Director — Sotio Biotech Inc.
Locations (16):
- Czechia (13):
  - Brno
  - Hradec Králové
  - Jindřichův Hradec
  - Kutná Hora
  - Náchod
  - Olomouc
  - Ostrava
  - Pardubice
  - Pilsen
  - Prague
  - Příbram
  - Ústí nad Labem
  - Zlín
- Slovakia (3):
  - Košice
  - Piešťany
  - Poprad

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hensler M, Rakova J, Kasikova L, Lanickova T, Pasulka J, Holicek P, Hraska M, Hrnciarova T, Kadlecova P, Schoenenberger A, Sochorova K, Rozkova D, Sojka L, Drozenova J, Laco J, Horvath R, Podrazil M, Hongyan G, Brtnicky T, Halaska MJ, Rob L, Ryska A, Coosemans A, Vergote I, Garg AD, Cibula D, Bartunkova J, Spisek R, Fucikova J. Peripheral gene signatures reveal distinct cancer patient immunotypes with therapeutic implications for autologous DC-based vaccines. Oncoimmunology. 2022 Jul 22;11(1):2101596. doi: 10.1080/2162402X.2022.2101596. eCollection 2022. PMID 35898703
- [Derived] Palata O, Podzimkova Hradilova N, Mysikova D, Kutna B, Mrazkova H, Lischke R, Spisek R, Adkins I. Detection of tumor antigens and tumor-antigen specific T cells in NSCLC patients: Correlation of the quality of T cell responses with NSCLC subtype. Immunol Lett. 2020 Mar;219:46-53. doi: 10.1016/j.imlet.2020.01.001. Epub 2020 Jan 10. PMID 31931024